CLINICAL TRIAL: NCT02399202
Title: A Phase I, Open-label, Multi-center, Single Dose, Parallel Group Study to Evaluate the Pharmacokinetics and Safety of LCI699 in Subjects With Varying Degrees of Impaired Renal Function Compared to Subjects With Normal Renal Function
Brief Title: A Phase I Study of Osilodrostat (LCI699) in Healthy Volunteers and Subjects With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCI699C2104; 2014-003528-35 (EudraCT Number)
Record Dates: First submitted 2015-03-20; First posted 2015-03-26 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-07

CONDITIONS: Renal Impairment
Keywords: Renal impairment, osilodrostat, LCI699
MeSH Terms: conditions — Renal Insufficiency | interventions — Osilodrostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osilodrostat ( LCI699) (Experimental): Each participant will undergo a 28 day screening /baseline period (day-28 to Day -1), followed by a 4 day treatment period ( a single 30 mg dose of LCI699 (Day 1) with 4 days of PK smple collection
  Interventions: Drug: osilodrostat

INTERVENTIONS:
Drug: osilodrostat

SUMMARY:
To characterize the pharmacokinetics of LCI699 following a single oral dose in adult subjects with various degrees of impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Weight must be ≥50 kg and BMI must be between 18-35 kg/m2
* Subjects must have stable renal disease without evidence of progressive decline in renal function (stable renal disease is defined as no significant change, such as, stable eGFR <90 mL/min, for 12 weeks prior to study entry) Other than renal impairment, subjects must be stable and appropriately managed relative to chronic diseases (such as diabetes and hypertension)

Exclusion Criteria:

* History of any surgical or medical condition other than renal impairment which might significantly alter the absorption, distribution, metabolism or excretion of drugs.
* Subjects with ongoing alcohol or drug abuse within 1 month prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Subjects with screening 12-lead ECG QTcF of > 450 msec for males or > 460 msec for female
* History of diabetes mellitus (Type 1 or 2) or blood glucose of >125 mg/dl at screening
* Subjects with potassium levels greater than the upper limit of normal (>ULN)

Other protocol defined Inclusion/Exclusion may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK in plasma) of a single dose of 30 mg osilodrostat: AUClast | Pre-dose (Day 0), and at timepoints 05.1,1.5,2,3,4,6,8,12,24,36,28 and 72 hours post dose
  To assess the influence of renal impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of renal impairment compared to subjects with normal renal function.
Pharmacokinetics (PK in plasma) of a single dose of 30 mg osilodrostat: AUCinf | Pre-dose (Day 0), and at timepoints 05.1,1.5,2,3,4,6,8,12,24,36,28 and 72 hours post dose
  To assess the influence of renal impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of renal impairment compared to subjects with normal renal function.
Pharmacokinetics (PK in plasma) of a single dose of 30 mg osilodrostat: Cmax | Pre-dose (Day 0), and at timepoints 05.1,1.5,2,3,4,6,8,12,24,36,28 and 72 hours post dose
  To assess the influence of renal impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of renal impairment compared to subjects with normal renal function.
Pharmacokinetics (PK in urine) of a single dose of 30 mg osilodrostat: CL/F | Pre-dose (Day 0), and at timepoints 05.1,1.5,2,3,4,6,8,12,24,36,28 and 72 hours post dose
  To assess the influence of renal impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of renal impairment compared to subjects with normal renal function.

SECONDARY OUTCOMES:
The relationship between PK parameters (, T1/2, V2/F and urine AeOt) | Pre-dose (Day 0), and at timepoints 05.1,1.5,2,3,4,6,8,12,24,36,28 and 72 hours post dose
Number of participants with adverse events | Pre-treatment, during treatment (Day1) and 30 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CLCI699C2104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16047